CLINICAL TRIAL: NCT00120952
Title: A Comparison Between Titanium Femoral Stem and Cobalt-Chromium Femoral Stem in Cemented Hip Arthroplasty. A Randomized Prospective Roentgen Stereogrammetric Analysis.
Brief Title: A Comparison Between Titanium Femoral Stem and Cobalt-Chromium Femoral Stem in Cemented Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-2351-02
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
Keywords: RSA; Osteoarthritis; Hip arthroplasty; DEXA; Titanium; Cobalt chromium; Bone cement
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: Bi-Metric femoral implant (titanium versus cobalt-chromium)

SUMMARY:
In this randomised study, the migration of a specific cemented titanium femoral stem will be compared with a similar cemented cobalt-chromium stem using Roentgen stereogrammetric analysis (RSA). In addition, the periprosthetic bone mineral density (BMD) will be evaluated to point out any interference from the modulus of the stem investigated.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip
* Spinal anesthesia
* Informed written consent

Exclusion Criteria:

* Neuromuscular disease in the affected leg
* Vascular disease in the affected leg
* Fracture sequelae in the affected hip
* Weight over 100 kg
* Regular non-steroid anti-inflammatory drug (NSAID) intake in the postoperative period

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2010-01

PRIMARY OUTCOMES:
Migration of femoral components evaluated by RSA

SECONDARY OUTCOMES:
Periprosthetic BMD changes evaluated by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, DMSc, Study Chair — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopaedic Department, Ribe County Hospital, Esbjerg, Denmark